CLINICAL TRIAL: NCT02180906
Title: Biomarkers in Necrotizing Soft Tissue Infections - Aspects of the Innate Immune Response
Brief Title: Biomarkers in Patients With Flesh-eating Bacterial Infections
Acronym: BIONEC
Status: Completed | Type: Observational
Sponsor: Ole Hyldegaard (Other)
Collaborators: Seventh Framework Programme (Other)
Responsible Party: Sponsor-Investigator, Ole Hyldegaard, Ole Hyldegaard, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: BIONEC1-MBH-2014
Record Dates: First submitted 2014-06-29; First posted 2014-07-03 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Necrotizing Soft Tissue Infection; Necrotizing Fasciitis; Gas Gangrene; Fournier Gangrene
Keywords: Fasciitis; Gangrene; Fasciitis, Necrotizing; Soft Tissue Infections; Fournier's Gangrene; Streptococcal septic shock syndrome; Flesh eating bacteria; Meleneys ulcer; Wounds and Injuries; Streptococcus pyogenes; Staphylococcus aureus; Immunopathogenesis; Soft Tissue Infections/blood; Necrosis/blood; Necrosis/diagnosis; Necrosis/mortality; Necrosis/surgery; Prognosis; Risk Factors; Bacterial Infections; Infection; Skin Diseases, Bacterial; Observational study; Biological markers
MeSH Terms: conditions — Fasciitis, Necrotizing; Gas Gangrene; Fournier Gangrene; Fasciitis; Gangrene; Soft Tissue Infections; Wounds and Injuries; Staphylococcal Infections; Necrosis; Disease; Bacterial Infections; Infections; Skin Diseases, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and plasma/serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with NSTI: Definition: An infection that requires acute hospitalization with intensive care treatment and/or surgery as a consequence of severe soft tissue infection in subcutis, muscle and/or fascia and are spreading along tissue structures.

SUMMARY:
The purpose of this study is to investigate the immune response in patients with necrotizing soft tissue infections (NSTI). The investigation will focus on inflammatory and vasoactive biomarkers as prognostic markers of severity and mortality at admission to Rigshospitalet and the following 3 days

DETAILED DESCRIPTION:
Necrotizing soft tissue infection (NSTI) is a complex, multi-factorial disease with diverse microbiological etiology and varying co-morbidities. The rapidly spreading infection may cause extensive soft tissue damage, limb loss, and multiple organ failure. The incidence of NSTIs has increased over the past years and the fatality rates are still high despite increased focus on these patients (20-30%). The extensive inflammatory response is thought to be a main course of death. However, it is unknown which biomarkers that are responsible for the deleterious effects and how these molecular mediators are modulated during the infection and treatment regimes. Thus, there is a need for novel insight into the immune system disturbances in order to improve outcome of NSTIs.

Location: Copenhagen University Hospital, Rigshospitalet, Denmark.

Design: Observational cohort study.

Cohort: NSTI patients in Denmark.

Controls: 50-100 Patients undergoing elective, orthopedic surgery at Rigshospitalet.

Biomarkers: The investigators will focus on three major groups of biomarkers: Acute-phase proteins, cytokines and vasoactive biomarkers.

Sample size calculations:

1. Acute-phase proteins: The investigators expect a mean PTX3-concentration at admission at 120 nmol/L in patients without septic shock and a mean PTX3-concentration at 210 nmol/L in patients with septic shock. With an estimated standard deviation at 100 nmol/L, the inclusion of 52 patients will be able to detect a significant difference with a statistical power of 90% at a 5% significance level. Since the groups are unequal the investigators will need to include 82 patients (N'=52(1+4)^2/4*4).
2. Cytokines: In a pilot study with seven NSTI patients, the investigators found a minimal clinically relevant difference in IL-6 concentration in NSTI patients with LRINEC < 6 and ≥ 6 to be 1050 pg/ml. With an estimated standard deviation at 2000 pg/ml, the inclusion of 114 patients will be able to detect a significant difference with a statistical power of 80% at a 5% significance level.
3. Vasoactive proteins: The investigators expect a mean NOx-concentration at admission at 90 μmol/L in patients without septic shock and a mean NOx-concentration at 145 μmol/Lin patients with septic shock. With an estimated standard deviation at 70 μmol/L, the inclusion of 70 patients will be able to detect a significant difference with a statistical power of 90% at a 5% significance level. Since the groups are unequal the investigators will need to include 110 patients (N'=70(1+4)^2/4*4).

Data: Data will be handled according to the National Data Protection Agency. All original records (incl. consent forms and questionnaires) will be archived at trial site for 15 years. The National Data Protection Agency has approved the biobank (2007-58-0015, J. nr. 30-1282).

Ethics: The trial will adhere to the Helsinki Declaration and Danish law. The National Ethics Committee and the Regional Ethics Committee have approved the inclusion of the NSTI patients (CVK-1211709) and the control patients, including biomarker analyses (H-2-2014-071).

Biomarker analyses, data extraction and interpretation will be performed once the recruiting of participants has ended.

ELIGIBILITY:
Inclusion Criteria for patients with NSTI:

* Necrotizing soft tissue infection based on surgical findings
* Age >18 years
* Admitted to/planned to be admitted to the ICU at Rigshospitalet and/or operated for NSTI at Rigshospitalet

Exclusion Criteria for patients with NSTI:

* Patients who at the operating theatre were categorized as non-NSTI patients

Inclusion Criteria for control patients:

* Patients undergoing elective orthopedic surgery (non-pathologic fractures, joint replacement surgery, back surgery) at Rigshospitalet
* Age >18 years

Exclusion Criteria for control patients:

* Patients with ongoing infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All NSTI patients treated at the University Hospital of Copenhagen, Rigshospitalet
Sampling Method: Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2013-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
PTX3, NOx and IL-6 as early markers of disease severity in NSTI patients with and without septic shock | Admission, first 24 hours
  Primary analysis: Association between PTX3-, NOx-, and IL6-concentration and septic shock (PTX3, NOx) or LRINEC ≥ 6 (IL-6) in NSTI patients at time of admission to Rigshospitalet

SECONDARY OUTCOMES:
Mortality | 28, 90, 180 days
Amputation rate | During ICU admission (expected average of 8 days)
  At any anatomical site
ICU-scoring systems | During ICU admission (expected average of 8 days)
  SAPS II (day 1) APACHE II (day 1) SOFA, GCS excluded (day 1-7), Anaya-score
Multiple organ failure | During ICU admission (expected average of 8 days)
Number of debridements | During ICU admission (expected average of 8 days)
Microbial etiology | During ICU admission (expected average of 8 days)
  Tissue and blood samples
Time from admission to primary hospital until first surgery/debridement | 2 days
Ventilator treatment, renal replacement therapy, vasopressor treatment during stay at ICU | During ICU admission (expected average of 8 days)
Steroid treatment (injection/oral intake) up to development of NSTI | Up to 7 days before surgical diagnose at primary hospital
Inflammatory biomarkers | Admission and the following 3 days
  Secondary analysis: The association between inflammatory biomarkers such as CRP, procalcitonin, mannose-binding-lectin and ficolin-1,2,3, cytokines and septic shock, LRINEC ≥ 6 and SAPS II at admission and the following 3 days
Vasoactive biomarkers | Admission and the following 3 days
  Secondary analysis: The association between vasoactive biomarkers such as NOx (nitrite, NO2-, and nitrate, NO3-,), L-arginine, asymmetric dimethylarginine, hydrogen sulfide, reactive oxygen species, ICAM-1, E-selectin and septic shock, LRINEC ≥ 6 and SAPS II at admission and the following 3 days
The effects of immunoglobulin on inflammatory biomarkers | Admission and the following 3 days
  A subgroup analysis will be performed on patients randomized to immunoglobulin or saline as immunoglobulin might affect the biomarker response (PTX3, NO, IL-6). The randomized double-blinded study was initiated April 2014 and registered at ClinicalTrials.gov (NCT02111161).
Biomarkers and Severity of disease | Admission and the following 3 days
  Subgroup analysis: Systemic inflammatory response syndrome, sepsis, severe sepsis and septic shock will be diagnosed according to standardized criteria (American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference Committee) and the biomarkers will be investigated to see if there is a correlation between disease severity and mortality in these groups.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bo Hansen, MD, Principal Investigator — Rigshospitalet, Denmark; Ole Hyldegaard, MD, PhD, Study Director — Rigshospitalet, Denmark
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hasham S, Matteucci P, Stanley PR, Hart NB. Necrotising fasciitis. BMJ. 2005 Apr 9;330(7495):830-3. doi: 10.1136/bmj.330.7495.830. PMID 15817551
- [Background] Sultan HY, Boyle AA, Sheppard N. Necrotising fasciitis. BMJ. 2012 Jul 20;345:e4274. doi: 10.1136/bmj.e4274. No abstract available. PMID 22822005
- [Background] Golger A, Ching S, Goldsmith CH, Pennie RA, Bain JR. Mortality in patients with necrotizing fasciitis. Plast Reconstr Surg. 2007 May;119(6):1803-1807. doi: 10.1097/01.prs.0000259040.71478.27. PMID 17440360
- [Background] Muller B, Peri G, Doni A, Torri V, Landmann R, Bottazzi B, Mantovani A. Circulating levels of the long pentraxin PTX3 correlate with severity of infection in critically ill patients. Crit Care Med. 2001 Jul;29(7):1404-7. doi: 10.1097/00003246-200107000-00017. PMID 11445697
- [Background] Bastrup-Birk S, Skjoedt MO, Munthe-Fog L, Strom JJ, Ma YJ, Garred P. Pentraxin-3 serum levels are associated with disease severity and mortality in patients with systemic inflammatory response syndrome. PLoS One. 2013 Sep 9;8(9):e73119. doi: 10.1371/journal.pone.0073119. eCollection 2013. PMID 24039869
- [Background] Panacek EA, Marshall JC, Albertson TE, Johnson DH, Johnson S, MacArthur RD, Miller M, Barchuk WT, Fischkoff S, Kaul M, Teoh L, Van Meter L, Daum L, Lemeshow S, Hicklin G, Doig C; Monoclonal Anti-TNF: a Randomized Controlled Sepsis Study Investigators. Efficacy and safety of the monoclonal anti-tumor necrosis factor antibody F(ab')2 fragment afelimomab in patients with severe sepsis and elevated interleukin-6 levels. Crit Care Med. 2004 Nov;32(11):2173-82. doi: 10.1097/01.ccm.0000145229.59014.6c. PMID 15640628
- [Background] Su YC, Chen HW, Hong YC, Chen CT, Hsiao CT, Chen IC. Laboratory risk indicator for necrotizing fasciitis score and the outcomes. ANZ J Surg. 2008 Nov;78(11):968-72. doi: 10.1111/j.1445-2197.2008.04713.x. PMID 18959694
- [Derived] Kristensen MK, Hansen MB, Madsen MB, Hansen CB, Pilely K, Hyldegaard O, Garred P. Complement Activation Is Associated With Mortality in Patients With Necrotizing Soft-Tissue Infections-A Prospective Observational Study. Front Immunol. 2020 Jan 31;11:17. doi: 10.3389/fimmu.2020.00017. eCollection 2020. PMID 32082310
- [Derived] Hansen MB, Rasmussen LS, Garred P, Bidstrup D, Madsen MB, Hyldegaard O. Pentraxin-3 as a marker of disease severity and risk of death in patients with necrotizing soft tissue infections: a nationwide, prospective, observational study. Crit Care. 2016 Feb 15;20:40. doi: 10.1186/s13054-016-1210-z. PMID 26880104
- [Derived] Hansen MB, Simonsen U, Garred P, Hyldegaard O. Biomarkers of necrotising soft tissue infections: aspects of the innate immune response and effects of hyperbaric oxygenation-the protocol of the prospective cohort BIONEC study. BMJ Open. 2015 May 11;5(5):e006995. doi: 10.1136/bmjopen-2014-006995. PMID 25967993
- See also: Research website: INFECT-study. Further description of funding from EU 7th Framework Programme — http://www.fp7infect.eu